CLINICAL TRIAL: NCT03743441
Title: A Double-blind Randomized Controlled Trial of Physiotherapy Treatment for Chronic Achilles Tendinopathy
Brief Title: Physiotherapy Treatment for Chronic Achilles Tendinopathy
Acronym: PhyCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Universidade do Vale do Paraíba (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20161107
Record Dates: First submitted 2018-11-06; First posted 2018-11-16 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Achilles Tendinopathy
Keywords: Chronic tendinopathy; Low-level Laser Therapy; LLLT; Photobiomodulation; Cryotherapy; Exercise therapy; Randomized Clinical Trial; RCT; Placebo-controlled
MeSH Terms: interventions — Low-Level Light Therapy; Exercise Therapy; Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two identical laser devices are used, where one is active and the other is sham. One laser device has a 3x60 mW output power and the other one has 0 mW output power (sham).
  These are labelled with yellow or blue tape by a secretary who is otherwise not participating in the study.
  Since the laser device has an invisible beam (904 nm wavelength) and is of such low power that heat is not detected, both the participant and the clinician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + Cryotherapy + LLLT (Active Comparator)
  Interventions: Other: Low-level Laser Therapy; Other: Exercise therapy; Other: Cryotherapy
- Exercise + Cryotherapy + Sham LLLT (Sham Comparator)
  Interventions: Other: Sham Low-level Laser Therapy; Other: Exercise therapy; Other: Cryotherapy

INTERVENTIONS:
Other: Low-level Laser Therapy — LLLT, 904 nm wavelength, 3 Joules per treatment point in accordance with World Association for Laser Therapy (WALT) guidelines.
  Other Names: Photobiomodulation
  Arms: Exercise + Cryotherapy + LLLT
Other: Sham Low-level Laser Therapy — Same procedure as in the LLLT group with the exception of laser irradiation (0 mW mean output power).
  Other Names: Sham Photobiomodulation
  Arms: Exercise + Cryotherapy + Sham LLLT
Other: Exercise therapy — Concentric and eccentric exercises with a total duration of approximately 20 minutes.
Other: Cryotherapy — Twenty minutes of cryotherapy applied to the Achilles tendon.

SUMMARY:
Laser treatment with the proper dosage has been found effective in the treatment of chronic Achilles tendinopathy, and animal research indicate that a combination of cryotherapy followed by LLLT could yield an even better result.

Thus, the main purpose of this project is to test if the addition of low level laser therapy can enhance the treatment result of exercise and cryotherapy in patients with chronic Achilles tendinopathy, yielding less pain and higher function.

ELIGIBILITY:
Inclusion Criteria:

* Achilles tendinopathy with a minimum duration of three months, pathological appearance of the Achilles tendon with thickened tendon and structural changes of the tendons matrix.

Exclusion Criteria:

* Cortisone injection within the last 6 months, systemic inflammatory disease, previous suture/surgery of the Achilles tendon, pregnancy or familial hypercholesterolemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
The VISA-A questionnaire: An index of the severity of Achilles tendinopathy | Change from baseline to week 4 and 12
  Range 0-100
Pain (Numerical Rating Scale) | Change from baseline to week 4 and 12
  Range 0-10

SECONDARY OUTCOMES:
Pain pressure threshold algometry | Change from baseline to week 4 and 12
  Algometer placed upon the Achilles tendon at the most sensitive spot identified by palpation. If it is unclear what the most sensitive spot is, the algometer is placed 2 cm proximal from the calcaneus.
Palpation tenderness | Change from baseline to week 4 and 12
  The Achilles tendon is palpated by the assessor while the participant is lying prone. The participant indicates whether the pressure produces pain by answering yes/no.
Single legged heel raise | Change from baseline to week 4 and 12
  The participant stands solely on one leg and lifts the heel of the floor. The distance from the heel to the floor is measured.
Jump for distance | Change from baseline to week 4 and 12
  One leg take-off and landing
Thickness of the Achilles tendon | Change from baseline to week 4 and 12
  Measured with real time ultrasonography in a longitudinal and sagittal view.
Neovascularization in the Achilles tendon | Change from baseline to week 4 and 12
  Doppler activity measured with real time ultrasonography in a longitudinal and sagittal view.
Qualitative assessment of structural changes of the Achilles tendon | Change from baseline to week 4 and 12
  Structural changes are assessed by real time ultrasonography. The structural changes of the Achilles tendon is scored as absent, mild, moderate, or severe.
Qualitative assessment of effusion within of the Achilles tendon | Change from baseline to week 4 and 12
  Amount of effusion is assessed by real time ultrasonography. The amount of effusion within and around the Achilles tendon is scored as absent, mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Ingvill F Naterstad, MSc, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No